CLINICAL TRIAL: NCT05114070
Title: Build a Decision Aid Tool to Help Emergency Intensive Care Specialists in the Context of Hypoxic Ischemic Encephalopathy. NEWBORN NEURO-DIGITAL STUDY
Brief Title: Build a Decision Aid Tool to Help Emergency Intensive Care Specialists in the Context of Hypoxic Ischemic Encephalopathy
Acronym: NewbornDS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 210070
Record Dates: First submitted 2021-07-09; First posted 2021-11-09 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Encephalopathy
Keywords: Full Term Newborn; EEG; HIE
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Decision of hypothermia — Decision of hypothermia thanks to EEG signal

SUMMARY:
The project aims at designing a machine learning solution able to recognize characteristics signals patterns of brain damages in full term babies born within a context of Hypoxic Ischemic Encephalopathy (HIE)

DETAILED DESCRIPTION:
Retrospective study based on a digital EEG signal library intending to design, train and test an efficient AI solution for hypothermia protocol start indications.

The output of the Project is to make available to pediatric resuscitation units an adequate tool to guide them in the decision of hypothermia protocol start in a general context of neurophysiologist competence scarcity. EEG signal that would allow the algorithm design will be based on several parameters of the conventional EEG and not only on signal amplitude

ELIGIBILITY:
Inclusion Criteria:

* Full term (> 36 weeks)
* HIE context
* EEG recording before 6 hours of life

Exclusion Criteria:

-Opposition of parental authority holders of a patient born after 2015

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies born within a context of HIE (Hypoxic Ischemic Encephalopathy)
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Decision of hypothermia protocol start | 6 months
  Use of EEG signal in order to develop an algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital TROUSSEAU, Paris, France

REFERENCES:
- [Derived] Fiammante M, Vermersch AI, Vidailhet M, Chavez M. A simple EEG-based tool to guide therapeutic hypothermia decisions in neonatal hypoxic-ischemic encephalopathy. Comput Methods Programs Biomed. 2026 Feb 1;274:109166. doi: 10.1016/j.cmpb.2025.109166. Epub 2025 Nov 13. PMID 41260106